CLINICAL TRIAL: NCT00778167
Title: A Phase I/Randomized Phase II Study of the Anti-IGF-1R Monoclonal Antibody IMC-A12 in Combination With Erlotinib Compared With Erlotinib Alone in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Erlotinib Hydrochloride With or Without Cixutumumab in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00286; NCI-2009-00286 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000617094; UCHSC-08-0044; COMIRB 08-0044 (Other: University of Colorado at Denver); 8148 (Other: CTEP); P30CA046934 (NIH); N01CM62209 (NIH); R21CA135595 (NIH)
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2013-03

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cixutumumab; Erlotinib Hydrochloride

ARMS (2):
- Arm I (Enzyme inhibitor therapy) (Experimental): Patients receive erlotinib hydrochloride PO once daily on days 1-21. Patients with documented disease progression may cross over and receive treatment on arm II.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis
- Arm II (Enzyme inhibitor and monoclonal antibody therapy) (Experimental): Patients receive erlotinib hydrochloride PO as in arm I and cixutumumab IV over 1 hour on days 1, 8, and 15.
  Interventions: Biological: cixutumumab; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cixutumumab — Given IV
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
  Arms: Arm II (Enzyme inhibitor and monoclonal antibody therapy)
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I/II trial is studying the side effects and best dose of cixutumumab and to see how well erlotinib hydrochloride works when given together with or without cixutumumab in treating patients with stage III or stage IV non-small cell lung cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether erlotinib hydrochloride is more effective when given together with or without cixutumumab in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a tolerable dose of IMC-A12 (cixutumumab) in combination with erlotinib (erlotinib hydrochloride) in the target NSCLC population to be administered in the randomized phase II study section.

II. To determine the difference in PFS between the anti-IGF-1R monoclonal antibody IMC-A12 in combination with erlotinib compared to erlotinib alone in the target NSCLC population.

SECONDARY OBJECTIVES:

I. To evaluate the safety, tolerability, and adverse event profile of IMC-A12 in combination with erlotinib in patients with advanced non-small cell lung cancer.

II. To describe preliminary evidence of clinical activity of the combination of IMC-A12 and erlotinib.

III. To determine the difference in overall response rate (ORR) between the two treatment arms.

IV. To determine the response duration in patients who achieve an objective response in either study arm.

V. To describe the response rate, time to disease progression, and response duration in the population who cross over to the combination arm after disease progression with single agent erlotinib therapy.

TERTIARY OBJECTIVES:

I. To explore the prognostic/predictive significance of the immunohistochemical, mutational, and cytogenetic profiles from archived tumor tissue of key elements of the EGFR, IGF-1R and other relevant signaling pathways in relationship to clinical benefit from treated individuals in both Part A and Part B sections of the study.

II. To explore the prognostic/predictive significance of serum circulating markers (ligands and binding proteins) and serum proteomic profiles pre-treatment and at progression in both Part A and Part B sections of the study.

III. To explore the impact of SNPs in germline and tumor derived DNA on toxicity and anti-cancer activity within both Part A and Part B sections of the study.

IV. To explore the impact of SNPs in germline DNA on erlotinib pharmacokinetics within both Part A and Part B sections of the study.

OUTLINE: This is a multicenter study that includes a single-arm safety evaluation phase I followed by a randomized phase II study.

Initially, patients are enrolled in the safety evaluation phase. If ≤ 2 of 10 patients experience a dose-limiting toxicity, then the study may proceed to the randomized phase. Safety evaluation phase I: Patients receive cixutumumab intravenously (IV) over 1 hour on days 1, 8, 15, and 22 and erlotinib hydrochloride orally (PO) once daily on days 1-28. Courses repeat every 28 days until disease progression or unacceptable toxicity.

Randomized phase II: Patients are stratified according to performance status, history of smoking (never vs ex vs current), stage of disease (IIIA vs IIIB without malignant effusion vs IIIB with malignant effusion vs IV), EGFR mutation (present vs absent vs not known), and disease histology (squamous vs non-squamous). Patients are randomized to 1 of 2 treatment arms.

ARM 1: Patients receive erlotinib hydrochloride PO once daily on days 1-21. Patients with documented disease progression may cross over and receive treatment on arm II.

ARM II: Patients receive erlotinib hydrochloride PO as in arm I and cixutumumab IV over 1 hour on days 1, 8, and 15. Patients receive treatment in both arms as in the safety evaluation portion. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Archived tissue and blood samples are collected periodically for pharmacokinetic analysis of erlotinib hydrochloride; pharmacogenomic analysis of EGRF, IGF1R, and CYP3A4/5 mutations; IHC and FISH analysis of IGF1R, EGFR, cMET, ras, Akt1, and EMT; proteomic analysis of serum ligand/binding proteins (i.e., IGF1, IGF2, IGFBPs, EGF, HRG, and TGF-α) using matrix-assisted laser desorption/ionization time of flight mass spectrometry (MALDI-TOF); mutational status analysis of EGFR and related pathway proteins; and RT-PCR analysis.

After completion of study therapy, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIA, IIIB, or IV disease
  * Mixed histology permitted provided small-cell elements are not present
* Measurable disease, defined as ≥ 1unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have failed ≥ 1 platinum-containing chemotherapy regimen
* CNS metastases are eligible if received prior radiotherapy to site(s) of CNS metastatic disease, or have had definitive resection of CNS metastatic disease and have no overt evidence of neurological deficits, are not requiring anti-epileptics, remain asymptomatic, and have been off steroids for ≥ 8 weeks
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* Leukocytes ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 100,000/mm³
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Fasting serum glucose < 120 mg/dL OR normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to anti-IGF-1R recombinant monoclonal antibody IMC-A122 or erlotinib hydrochloride
* No poorly controlled diabetes mellitus

  * Patients with a history of diabetes mellitus are eligible, provided their blood glucose is within normal range at screening and they are on a stable dietary or therapeutic regimen for this condition
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No inability to take oral medications or, in the investigator's opinion, gastrointestinal conditions or abnormalities likely to influence the absorption of oral medications
* No prior or concurrent exposure to other EGFR or IGFR inhibitors
* Recovered from all prior therapy with acute effects resolved to ≤ grade 1
* At least 28 days since prior anticancer or investigational agent (within predicted 5 half-lives of agent)
* More than 4 weeks since prior radiotherapy to target lesions and documented disease progression at these sites
* More than 2 weeks since prior radiotherapy to non-target lesions
* More than 4 months since prior major surgery or hormonal therapy (other than replacement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Camidge, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado, Denver, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2008 and October 2010, 18 patients were enrolled across cohorts 1 to 3.
Pre-assignment Details: Phase I of the study, determining a tolerable dose of IMC-A12 in combination with erlotinib, was completed. Because of concerns about the achievable dose intensity at the maximum tolerated dose, a randomized phase II study that would have involved Arm I in comparing full-dose erlotinib with the IMC-A12 in combination with erlotinib was cancelled.
Groups:
- Cohort 1: Cohort 1: Patients received oral erlotinib hydrochloride 150 mg once daily with cixutumumab 6 mg/kg IV on days 1, 8, 15, and 22 in 28-day cycles.
- Cohort 2: Cohort 2: Patients received oral erlotinib hydrochloride 150 mg once daily with cixutumumab 5 mg/kg IV on days 1, 8, 15, and 22 in 28-day cycles.
- Cohort 3: Cohort 3: Patients received oral erlotinib hydrochloride 150 mg once daily with cixutumumab 15 mg/kg IV in 21-day cycles.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 6 | 8 | 4
Completed | 6 | 8 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Patients received oral erlotinib hydrochloride 150 mg once daily with cixutumumab 6 mg/kg IV on days 1, 8, 15, and 22 in 28-day cycles.
- Cohort 2: Patients received oral erlotinib hydrochloride 150 mg once daily with cixutumumab 5 mg/kg IV on days 1, 8, 15, and 22 in 28-day cycles.
- Cohort 3: Patients received oral erlotinib hydrochloride 150 mg once daily with cixutumumab 15 mg/kg IV in 21-day cycles.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 6 | 8 | 4 | 18
Age, Customized [Number; unit: participants]
  <=48 years | 0 | 0 | 0 | 0
  Between 48 and 77 years | 6 | 8 | 4 | 18
  >=77 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 2 | 10
  Male | 4 | 2 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of IMC-A12 in Combination With Erlotinib Hydrochloride as Graded by Common Terminology Criteria for Adverse Event (CTCAE) Version 3.0 (DLTs During Cycle One)
Description: Patients were evaluable for cohort dose escalation/de-escalation decision making either if they experienced DLTs in cycle 1 or if they had completed 24 of the planned 28 days (85%) dosing of erlotinib and three of the four planned days of weekly dosing of cixutumumab (75%) in cycle 1 in cohorts 1 and 2 in the absence of DLTs. In cohort 3, patients were evaluable for tolerability if they had completed 18 days (85%) dosing of erlotinib and had received the planned day 1 dose of cixutumumab.
Time Frame: From time of first dose up to 28 days
Population: Patients were evaluated with history, physical examination, vital signs, and blood tests weekly through cycle 1 and on day 1 of each subsequent cycle. Incidence and severity of AEs were collected at each study visit and graded according to National Cancer Institute Common Toxicity Criteria for Adverse Events version 3.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 6 | 8 | 4
Participants | 4 | 1 | 2

ADVERSE EVENTS:
Time Frame: Weekly through cycle 1 and on day 1 of each subsequent cycle
Description: Patients were evaluated with history, physical examination, vital signs, and blood tests weekly through cycle 1 and on day 1 of each subsequent cycle. Incidence and severity of AEs were collected at each study visit
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=8) | Cohort 3 (N=4)
Fatigue (General disorders) | 5 (5) | 5 (5) | 3 (3)
Acneiform rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3)
Anorexia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Mucositis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Taste alteration (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Phase I of the study was completed but because of concerns about the achievable dose intensity at the maximum tolerated dose (MTD), the expansion into a randomized phase II study comparing full-dose erlotinib with the combination was cancelled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less